CLINICAL TRIAL: NCT02769312
Title: Pilot Testing of Theta-Burst Neuromodulation for Chronic PTSD
Brief Title: Theta-Burst Neuromodulation for PTSD
Acronym: TBS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2032-P; I21RX RX002032 (Other Grant/Funding Number: VA)
Record Dates: First submitted 2016-04-29; First posted 2016-05-11 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Chronic Post-Traumatic Stress Disorder
Keywords: Quality of Life; Post-Traumatic Stress Disorder; Transcranial Magnetic Stimulation; Feasibility studies
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham Stimulation (Sham Comparator): A sham coil is being used to compare against active coil.
  Interventions: Device: Sham stimulation
- Active Stimulation (Active Comparator): An active coil is being used to compare against sham coil.
  Interventions: Device: Theta burst stimulation

INTERVENTIONS:
Device: Theta burst stimulation — Theta burst transcranial magnetic stimulation
  Arms: Active Stimulation
Device: Sham stimulation — Sham Theta burst transcranial magnetic stimulation
  Arms: Sham Stimulation

SUMMARY:
The purpose of the proposed study is to evaluate initial feasibility and efficacy of Theta Burst Transcranial Magnetic Stimulation (TBS) as an adjunct treatment for Veterans with PTSD. Primary outcomes measures include a feasibility of TBS procedures, with secondary outcome measures focusing on changes in PTSD symptom severity and quality of life and social/occupation functioning.

DETAILED DESCRIPTION:
The purpose of the proposed study is to evaluate the feasibility of theta burst transcranial magnetic stimulation (TBS) as an adjunct treatment for Veterans with PTSD. This project will result in development of methods needed to conduct an adequately powered, randomized controlled study of TBS for PTSD, which will assess the relationship between change in symptoms and quality of life. It will also lay the foundation for subsequent rehabilitation studies combining neuromodulation and psychotherapy in the longer term.

TBS has several advantages compared to standard repetitive Transcranial Magnetic Stimulation (rTMS), including its ability to deliver large numbers of stimulation pulses in a shorter time period, and a stimulation pattern that may specifically affect key brain regions involved in PTSD. The significance of this research is the development of a novel, non-invasive brain stimulation approach for PTSD recovery. This project will provide the foundation for the development of methods needed to conduct an adequately powered, randomized controlled study of TBS for PTSD to ultimately develop brain stimulation techniques that can be combined with evidence-based psychotherapy, to develop a more powerful, individualized rehabilitation option for Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic PTSD according to DSM-5 criteria
* Veteran (male or female)
* age between 18-70 years
* clinically symptomatic despite ongoing stable treatment regimens for at least 6 weeks prior to study procedures
* capable of independently reading and understanding patient information materials and providing informed consent

Exclusion Criteria:

* Cardiac pacemaker
* implanted device (deep brain stimulation) or metal in the brain
* cervical spinal cord
* or upper thoracic spinal cord
* pregnancy/lactation, or planning to become pregnant during the study
* lifetime history of moderate or severe traumatic brain injury (TBI)
* current unstable medical conditions
* current (or past if appropriate) significant neurological disorder, or lifetime history of:

  * seizure disorder
  * primary or secondary CNS tumors
  * stroke
  * cerebral aneurysm
  * primary psychotic disorder
  * bipolar I disorder
  * active moderate/severe substance use disorders (within the last month, excluding nicotine/caffeine
  * active suicidal intent or plan

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah S. Philip, MD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Philip NS, Barredo J, Aiken E, Larson V, Jones RN, Shea MT, Greenberg BD, van 't Wout-Frank M. Theta-Burst Transcranial Magnetic Stimulation for Posttraumatic Stress Disorder. Am J Psychiatry. 2019 Nov 1;176(11):939-948. doi: 10.1176/appi.ajp.2019.18101160. Epub 2019 Jun 24. PMID 31230462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants consented at a formal in-person eligibility determination (screening).
  Location: Providence, RI
Pre-assignment Details: 6 participants were excluded during pre-assignment.
  * 2 Not Eligible (1 due to the absence of Criterion A trauma, 1 declined to complete eligibility procedures)
  * 2 Withdrew Consent
  * 2 Discontinued (1 lost/unable to contact, 1 inpatient admission)
Groups:
- Sham Stimulation: Participants allocated to receive sham TBS during the double-blind period
- Active Stimulation: Participants allocated to receive active TBS during the double-blind period.
Period: Double-Blind (0-2 Weeks)
Arm/Group | Sham Stimulation | Active Stimulation
Started | 25 | 25
Completed | 23 | 24
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 0
Period: Unblinded (Optional 2-4 Weeks)
Arm/Group | Sham Stimulation | Active Stimulation
Started (Optional unblinded period. All participants received 2 weeks of active stimulation.) | 21 (2 participants chose not to continue with the unblinded period.) | 24
Completed | 20 | 23
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Follow-up
Arm/Group | Sham Stimulation | Active Stimulation
Started (1 month following the end of intervention.) | 23 | 24
Completed (Participants did not have to complete the unblinded period to complete the follow-up period.) | 22 | 23
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Stimulation | Active Stimulation | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 22 | 41
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12) | 49 (13) | 51 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 22 | 20 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 20 | 22 | 42
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50
Education [Count of Participants; unit: Participants]
  Less than high school | 1 | 1 | 2
  High school or equivalent | 5 | 2 | 7
  Some college | 7 | 11 | 18
  Trade or vocational degree | 0 | 3 | 3
  Bachelor's degree | 8 | 2 | 10
  Advanced degree and/or education beyond college | 3 | 2 | 5
  Multiple selections | 1 | 4 | 5
Employment Status [Count of Participants; unit: Participants]
  Full time | 4 | 6 | 10
  Part time | 2 | 1 | 3
  Unemployed | 9 | 10 | 19
  Retired | 9 | 6 | 15
  Multiple selections | 1 | 2 | 3
Military History [Count of Participants; unit: Participants] — Military Branch corresponding with participant's report of service branch at time of discharge.
  Participants
    Army | 8 | 8 | 16
    Navy | 6 | 8 | 14
    Marines | 1 | 2 | 3
    Air Force | 3 | 0 | 3
    No response | 7 | 7 | 14
Psychiatric Comorbidity [Count of Participants; unit: Participants]
  Major Depressive Disorder (MDD) | 25 | 25 | 50
  Bipolar II, most recent episode depressed | 3 | 2 | 5
  Substance Use Disorder (Mild) | 11 | 16 | 27
  Opoiod use disorder | 5 | 6 | 11
Prior Brain Stimulation [Count of Participants; unit: Participants]
  Transcranial Magnetic Stimulation | 2 | 0 | 2
  Electroconvulsive Therapy | 1 | 2 | 3
Mild Traumatic Brain Injury [Count of Participants; unit: Participants] | 5 | 7 | 12
Psychiatric History [Count of Participants; unit: Participants]
  Suicide attempt(s) | 6 | 6 | 12
  Inpatient hospitalization(s) | 15 | 13 | 28
PTSD Symptom Severity [Mean (Standard Deviation); unit: score on a scale] — CAPS-5, Clinician Administered PTSD Scale for DSM-5: structured interview to assess PTSD symptoms over the past month, items rated 0 = 'absent' to 4 = 'extreme/incapacitating,' total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms.
  PCL-5, PTSD Checklist for DSM-5: a 20-item self-report measure where participants are asked to respond about experience(s) "over past month,", items are rated 0 = "not at all bothered by" to 4 = "extremely bothered," total symptom severity score ranges 0-80, higher scores indicate more severe PTSD symptoms.
  score on a scale
    CAPS-5 Score | 47.36 (10.62) | 47.92 (9.97) | 47.64 (10.20)
    PCL-5 Score | 49.96 (11.37) | 49.40 (9.35) | 49.68 (10.31)
Social/Occupational Function & Quality of Life [Mean (Standard Deviation); unit: score on a scale] — SOFAS, Social and Occupational Function Scale: Clinician rating of social & occupational functioning. Scale of 0-100 with higher scores indicating higher functioning.
  QLESQ (General Quality of Life Index), Quality of Life Enjoyment and Satisfaction: A self-report scale covering multiple domains (physical health, subjective feelings, leisure time activities, social relationships, treatment) The General Quality of Life Index took the mean of all domains. Scores range from 0-5, with higher scores indicating higher quality of life.
  score on a scale
    SOFAS Score | 44.56 (14.94) | 44.32 (13.14) | 44.44 (13.92)
    QLESQ (General Quality of Life Index) | 2.57 (0.70) | 2.53 (0.75) | 2.55 (0.72)
Depressive Symptom Severity [Mean (Standard Deviation); unit: score on a scale] — IDSSR Score, Inventory of Depressive Symptomatology, Self-Report: participant self report of depressive symptoms over the past week based on 30 items (28 are scored), items rated 0-3. The total score can range from 0-84, with 0 being no depressive symptoms and 84 being severe depressive symptoms.
  score on a scale | 39.20 (11.52) | 42.84 (11.91) | 41.02 (11.74)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Retained, a Measure of Acceptability of TBS Procedures
Description: Measurement of TBS acceptability, measured using participant retention rates (all-cause discontinuation)
Time Frame: 2 weeks
Population: Data was analyzed in an intent-to-treat fashion, defined as participants that were randomized and received at least one iTBS session.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Stimulation | Active Stimulation
Number analyzed (Participants) | 25 | 25
Participants | 23 | 24

2. Secondary Outcome: Change in Quality of Life Due to TBS Treatment
Description: Change in the quality of life, using the quality of life questionnaire QLESQ - Quality of Life Enjoyment and Satisfaction Questionnaire (General Quality of Life Index).
  A self-report scale covering multiple domains (physical health, subjective feelings, leisure time activities, social relationships, treatment satisfaction) The General Quality of Life Index took the mean of all domains. Scores range from 0-5, with higher scores indicating higher quality of life.
Time Frame: Baseline and end of double-blind period (2 weeks)
Population: Data was analyzed in an intent-to-treat fashion. Primary outcomes were measured using analysis of variance to compare groups at the end of the 2-week double blind phase. Missing data was addressed using multiple imputation, with 20 imputations or maximum likelihood parameter estimation in mixed model analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Stimulation | Active Stimulation
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 2.57 (0.70) | 2.53 (0.75)
  End of Double-Blind | 2.71 (0.80) | 2.81 (0.78)
Statistical Analysis 1: Comparison: Sham Stimulation vs Active Stimulation; Test type: Other; p = 0.46, ANCOVA; Effect size (cohen's d) = 0.16

3. Secondary Outcome: Change in PTSD Symptom Severity
Description: Change in PTSD symptoms measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5).
  The CAPS-5 is a structured interview to measure for PTSD symptom change and presence/absence of PTSD, items rated 0 = 'absent' to 4 = 'extreme/incapacitating,' total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. Higher scores indicate more severe PTSD symptoms.
Time Frame: Baseline and end of double-blind period (2 weeks)
Population: Included all subjects who were randomized. Primary outcomes were measured using analysis of variance to compare groups at the end of the 2-week double blind phase. Missing data was addressed using multiple imputation, with 20 imputations or maximum likelihood parameter estimation in mixed model analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Stimulation | Active Stimulation
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 47.36 (10.62) | 47.92 (9.97)
  End of Double-Blind | 39.38 (13.77) | 38.58 (11.42)
Statistical Analysis 1: Comparison: Sham Stimulation vs Active Stimulation; Test type: Superiority; p = 0.61, ANCOVA; Effect size (cohen's d) = 0.12

4. Secondary Outcome: Change in Social/Occupational Functioning (QOL/SOF) Due to TBS Treatment
Description: Change measured using the social/occupational functioning assessment scale (SOFAS).
  Clinician rating of social & occupational functioning. Scale of 0-100 with higher scores indicating higher functioning.
Time Frame: Baseline and end of double-blind period (2 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Stimulation | Active Stimulation
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 44.56 (14.94) | 44.32 (13.14)
  End of Double-Blind | 48.08 (17.70) | 53.38 (16.96)
Statistical Analysis 1: Comparison: Sham Stimulation vs Active Stimulation; Test type: Superiority; p = .04, ANCOVA; Effect size (cohen's d) = 0.39

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the participants' study participation. Collection started the day the participant was consented and continued up to 1 month following the last treatment visit.
Groups:
- Pre-Allocation: Participants consented at formal in-person eligibility determination.
Arm/Group | Pre-Allocation | Sham Stimulation | Active Stimulation
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/56 | 2/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/56 | 2/25 | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Allocation (N=56) | Sham Stimulation (N=25) | Active Stimulation (N=25)
Inpatient hospitalization (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Allocation (N=56) | Sham Stimulation (N=25) | Active Stimulation (N=25)
Treatment site discomfort (Psychiatric disorders) | 0 (0) | 0 (0) | 6 (6)
Headache (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT02769312/Prot_SAP_000.pdf